CLINICAL TRIAL: NCT00784706
Title: Effect of Combined Therapy on Neglect Syndrome in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97-1391B
Record Dates: First submitted 2008-10-30; First posted 2008-11-04 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-07

CONDITIONS: Cerebrovascular Accidents
Keywords: stroke rehabilitation; perceptual deficits; kinematic analysis
MeSH Terms: conditions — Stroke | interventions — serum P-component; Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CIT with eye-patching (Experimental): The CIT addressed forced use of the affected UE and restricted the unaffected UE during training. Shaping skills were delivered while participants were forced to use their affected UE in the mass practice of functional tasks, such as drinking water and opening a jar. Participants wore a mitt on their unaffected hand and wrist for 6 hours/day during the 3-week training and reported their compliance in a daily log. Participants were also asked to wear glasses with a patch on the right lens to block the visual stimuli from the right side and force them to receive the stimuli from the left-side visual field.
  Interventions: Other: EP; Other: CIT
- constraint-induced therapy (Experimental): The intervention in this group resembled the intervention of the CIT+EP group, except participants did not wear the EP glasses.
  Interventions: Other: CIT
- conventional therapy (Active Comparator): traditional occupational therapy matched in intensity and duration with the other groups. The training program included stretching and weight bearing of the affected UE, improving the range of motion of the affected UE, muscle strengthening, and the practice of tasks used for functional training might involve the unaffected UE to assist in the affected UE; for example, stabilizing a bottle while opening its lid or moving pegs into holes on a board.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: EP — Participants were asked to wear glasses with a patch on the right lens to block the visual stimuli from the right side and force them to receive the stimuli from the left-side visual field.
  Other Names: eye-patching therapy
  Arms: CIT with eye-patching
Other: CIT — The CIT addressed forced use of the affected UE and restricted the unaffected UE during training. Shaping skills were delivered while participants were forced to use their affected UE in the mass practice of functional tasks, such as drinking water and opening a jar. Participants wore a mitt on their unaffected hand and wrist for 6 hours/day during the 3-week training and reported their compliance in a daily log.
  Other Names: constraint-induced therapy(CIT)
  Arms: CIT with eye-patching; constraint-induced therapy
Other: conventional therapy — Traditional occupational therapy matched in intensity and duration with the other groups. The training program included stretching and weight bearing of the affected UE, improving the range of motion of the affected UE, muscle strengthening, and the practice of tasks used for functional training might involve the unaffected UE to assist in the affected UE; for example, stabilizing a bottle while opening its lid or moving pegs into holes on a board.
  Arms: conventional therapy

SUMMARY:
The purpose of the current study is to evaluate motor and neglect recovery of stroke patients produced by CIT using kinematic and oculomotor assessment, together with conventional clinical measures.

DETAILED DESCRIPTION:
This project will be carried out using a short term constraint and training protocol targeting at subacute and chronic patients with motor and perceptual deficits. The outcome measures will include kinematic and oculomotor analyses, which have not been employed yet.

ELIGIBILITY:
Inclusion Criteria:

* a clinical cerebrovascular of right cerebral accident patients
* the age over 18-year-old
* demonstration of Brunnstrom stage III of the affected upper extremity
* patients with perceptual deficits
* no severe cognitive disorder, could understand and follow orders
* no severe equilibrium problems which will influence the intervention

Exclusion Criteria:

* recurrent of the stroke or epilepsy during the intervention
* patients with the neurological or psychical history, for example, alcoholism, drug poisoning or bipolar disorder
* injected the Botox into the affected upper extremity during the past 6 months
* participate in the other interventional study in the same time
* refuse subscribed the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Catherine Bergego Scale (CBS) | 2008-2009
  The CBS is a therapist-designed checklist to examine the effect of neglect syndrome on a patient's daily function in 10 real-life situations, such as grooming, dressing, or maneuvering a wheelchair. A 4-point scale is used in each item, ranging from 0 (no neglect) to 3 (severe neglect). Patients with a total score of 0 were considered as having no neglect in performing daily activities.

SECONDARY OUTCOMES:
Clinical measures at the impairment, activity, participation levels | 2008-2009
Eye movement analysis | 2008-2009
  An eye tracker system (Tobii 1750, with 1024 × 768 resolutions a 1 nd 30-Hz sampling rate) was used to record the participant's eye movement by detecting his or her pupil. To examine the possible improvement in abnormal eye movement after the intervention, the eye movement parameters included the fixation amplitude (the distance between the most left and the most right fixation points), the number of fixation points, and the fixation time in the left area (Left fixation points and Left fixation time). A fixation point is defined as the gaze point stays in 50 pixels on the screen over 30 ms and can be screened by a fixation filter function in the ClearView 2.0. A wider fixation amplitude, larger L fixation points, and longer L fixation time represent the alleviated syndrome of neglect.
kinematic variables | 2008-2009
  Kinematic analysis was used to detect UE and trunk movement. A 7-camera motion-analysis system (VICON MX; Oxford Metrics Inc., Oxford, UK)6 was linked to a personal computer to capture the movement of markers. Reference markers were placed on the seventh cervical vertebra (C7), the fourth thoracic vertebra (T4), the bilateral clavicles, midsternum, and the unaffected side of the acromion, middle of the humerus, lateral epicondyle,styloid process of the ulna and radius, and index nail. Kinematic variables included reaction time (second), normalized movement time (second), normalized total distance (mm), percentage of movement time where peak velocity (PPV) occurs, and trunk lateral shift.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-yi Wu, ScD, Principal Investigator — Department of Occupational Therapy, Chang Gung Univ.
Locations (1):
- Chang Gung Memorial Hospital, Kwei-shan, Toayuan County, Taiwan